CLINICAL TRIAL: NCT02697669
Title: The Role of Nuclear Imaging in Heart Failure: Correlation With Cardiac Function and Metabolism, Biomarkers and Clinical Prognosis
Brief Title: The Role of Nuclear Imaging in Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yen-Wen Wu, Chief of Cardiology Division of Cardiovascular Medical Center, Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: 101037_F
Record Dates: First submitted 2016-02-27; First posted 2016-03-03 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Heart Failure
Keywords: Heart failure; myocardial perfusion; single-photon emission tomography
MeSH Terms: conditions — Heart Failure | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 18F-FDG PET — Imaging
  Other Names: Imaging

SUMMARY:
Heart failure is a clinical syndrome of exercise intolerance and/or congestion. The potential roles of myocardial perfusion and metabolic abnormalities in subjects with cardiovascular risks, metabolic disease and heart failure assessed by nuclear dynamic imaging warrant further investigations. The study investigators propose that microvascular dysfunction and abnormal metabolic substrate shift precedes and triggers the onset of diastolic dysfunctions. The aims are (1) to develop and validate the noninvasive measurement of absolute myocardial blood flow (MBF) and myocardial flow reserve (MFR) by using dynamic imaging with a CZT camera, (2) to assess myocardial glucose metabolism by using 18F-FDG dynamic PET, and MBF, MFR and LV systolic and diastolic function by dynamic SPECT comprehensively in subjects at cardiovascular risks and metabolic disease, HFrEF and HFpEF, (3) to correlate with peripheral serum markers and blood mononuclear cells subsets with myocardial perfusion and metabolic abnormalities, and (4) to test the hypothesis of these imaging and blood markers in diagnosis and prognostic implications. The study investigators also assess myocardial metabolic utilization in healthy and mice model of different metabolic disorders (obesity, diabetes mellitus and hypertension) by using 18F-FDG dynamic micro PET/CT, as an in-vivo measures which could be used to better understanding the disease mechanism and evaluating therapeutic strategies.

DETAILED DESCRIPTION:
Heart failure (HF) is a clinical syndrome of exercise intolerance and/or congestion. The management of heart failure with reduced ejection fraction (HFrEF) has improved over the last decades. In contrast, little progress has been made in identifying evidence-based, effective treatments for heart failure with preserved ejection fraction (HFpEF, LVEF >50%). Treatments proven effective in HFrEF have failed to show significant benefit in patients with HFpEF. Potential contributors include an incomplete understanding of pathophysiology and poor matching of therapeutic mechanisms. The challenges of the use of diagnostic criteria, prognostic evaluation and treatment highlight the need for more research in this field.

This portion of HFpEF consists predominantly older age and high prevalence of co-morbidity such as overweight/obesity, diabetes mellitus, hyperlipidemia, metabolic syndrome and hypertension. The systemic pro-inflammatory state may induce coronary endothelial inflammation, microvasular dysfunction, myocardial substrate shift, myocardial and interstitial fibrosis that contribute to high diastolic left ventricular stiffness and HF development. Myocardial metabolic and perfusion imaging is a vital tool for understanding the physiologic consequences of HF. Absolute myocardial blood flow (MBF) and myocardial flow reserve (MFR) provide incremental diagnostic and prognostic information over relative perfusion alone. Recent development of dedicated cardiac SPECT cameras with better sensitivity and temporal resolution make dynamic SPECT imaging more practical. Quantitative 18F-FDG PET could be used as a means to measure myocardial metabolic changes. The study investigators propose that microvasular dysfunction and abnormal metabolic substrate shift precedes and triggers the onset of diastolic dysfunctions. The potential roles of myocardial perfusion and metabolic abnormalities in subjects with cardiovascular risks, metabolic disease and HFpEF assessed by nuclear dynamic imaging warrant further investigations.

The present project aims (1) to develop and validate the noninvasive measurement of absolute myocardial blood flow (MBF) and myocardial flow reserve (MFR) by using dynamic imaging with a CZT camera, (2) to assess myocardial glucose metabolism by using 18F-FDG dynamic PET, and MBF, MFR and LV systolic and diastolic function by dynamic SPECT comprehensively in participants at cardiovascular risks and metabolic disease, HFrEF and HFpEF, (3) to correlate with peripheral serum markers and blood mononuclear cells subsets with myocardial perfusion and metabolic abnormalities, and (4) to test the hypothesis of these imaging and blood markers in diagnosis and prognostic implications. The study investigators also assess myocardial metabolic utilization in healthy and mice model of different metabolic disorders (obesity, diabetes mellitus and hypertension) by using 18F-FDG dynamic micro PET/CT, as an in-vivo measures which could be used to better understanding the disease mechanism and evaluating therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Had a clinical diagnosis of heart failure and left ventricular systolic function (LVEF≤50%) or diastolic dysfunction who,
2. Clinical diagnosis of metabolic diseases (such as metabolic syndrome, obesity, diabetes, hyperlipidemia, microvascular diseases etc.), heart failure and high-risk groups.

Exclusion Criteria:

1. Important systemic disease (except for heart disease) such as cirrhosis, end-stage renal disease or active malignancy were estimated life expectancy of less than three months.
2. pregnant or lactating women.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Had a clinical diagnosis of heart failure and left ventricular systolic function (LVEF≤50%) or diastolic dysfunction who, or (2) Clinical diagnosis of metabolic diseases (such as metabolic syndrome, obesity, diabetes, hyperlipidemia, micro vascular diseases etc.), heart failure and high-risk groups.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
LV function | 12mo
  LVEF

SECONDARY OUTCOMES:
MACE | 5 years
  acute myocardial infarction, revasculiarization, ICD, heart transplantation, other cardiac surgery, hospitalization for heart failure, cardiac death, non-cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Wen Wu, MD, PhD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No